CLINICAL TRIAL: NCT07067177
Title: Prophylactic IV Paracetamol in Extremely Premature Infants
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ref#: Re11-06-024
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Patent Ductus Arteriosus in Preterm Infants; Patent Ductus Arteriosus After Premature Birth; Patent Ductus Arteriosus (PDA); Patent Ductus Arteriosus in Premature Infants
Keywords: Paracetamol prophylaxis; Paracetamol; Extremely premature infants; Extremely Premature; Neonates; Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Given prophylactic IV paracetamol (Active Comparator): The patients are given IV prophylactic paracetamol within the first 24 hours of life, first dose at the age of 6 hours, (15mg/kg/dose Q6hrs daily for five days).
  Interventions: Drug: Paracetamol (drug)
- No prophylactic paracetamol is given (No Intervention): No prophylactic paracetamol or placebo are given.

INTERVENTIONS:
Drug: Paracetamol (drug) — IV prophylactic paracetamol will be given prior to detection of PDA starting from 6 hours of age. It will be used to measure wethere this intervention reduces the risk of having persistant PDA, HsPDA, or any of their complications.
  Other Names: Acetaminophen; IV paracetamol
  Arms: Given prophylactic IV paracetamol

SUMMARY:
Purpose of the research Everyone is born with an opening between the chambers of the heart, called a ductus arteriosus. In most people, it closes on its own, but in infants born at less than 30 weeks or less than 1250 grams, there is a higher chance that it won't close on its own. So we give drugs to make it more likely that it closes. There are different medications that can do that, so we want to compare them to find which has the best effect.

Type of Research Intervention The drug will be given at age of 6 hours, then every 6 hours through IV.

Participant selection We are inviting suitable children with gestational age less than 30 weeks or birth weight less than 1250 grams.

Voluntary Participation Your participation in this research is entirely voluntary. It is your choice whether to participate or not. Whether you choose to participate or not, all the services you receive at this clinic will continue and nothing will change. If you choose not to participate in this research project, you will offered the treatment that is routinely offered in this hospital for the disease, and we will tell you more about it later. You may change your mind later and stop participating even if you agreed earlier.

The drug we want to give is paracetamol, it is a safe drug that has been tested on children of this age and proved to be safe. It has also been tested for this disease and shown to be effective. Some participants in the research will not be given this drug. Instead, they will be given Indomethacin, which is the most commonly used to prevent Ductus Arteriosus.

Procedures and Protocol

To compare the different medications, you will be randomly chosen as to whether you will receive which drug.

Standardly, different hospitals offer different treatments for the prevention of PDA. Some offer paracetamol, some offer indomethacin and some offer nothing. We will compare these options.

An echocardiography (imaging of the heart) will be done after 72 hours to check if the opening in the heart closed. In addition, close follow-up and attention will be given to check for its effects on the body. Lastly, blood tests will be taken at 24 hours, 72 hours, and after completing the course. They will measure liver enzymes in addition to others. A long-term follow-up will be done at 6 months.

B. Description of the Process

Duration The duration of the research will be for 6 months, but you will be asked to come back to the hospital after discharge only once after the 6 months.

Side Effects The medication is very unlikely to cause any side effects. However, the infant will be followed up closely to make sure that he doesn't develop any, and if he dose, we deal with it the right way and prevent it from harming the infant.

Risks By participating in this research, it is possible that your disease will not get better and that the new medicine won't work even as well as the old one. In this case, we have other medications that can be given to close it and solve the problem.

Benefits Your participation in this research will be of great benefit to the people and to other preterm infants. It will help us find out which medication is the best and give it to the upcoming newborns that are born early, like your child. Improving their lives.

Confidentiality The information that we collect from this research will remain confidential. Your child's name, condition, or research participation won't be discussed or released. The data will be stored in a safe place that isn't accessible except by a few people, then his data will be included among all others without mentioning his name or anything that may be used to identify him.

Sharing the Results After collection and analyzing the data, encoding it and removing all confidential information, the data of all the participants will be assembled into a scientific article and published in a scientific journal to help and reach more people. You will also be notified of the research outcomes before the paper.

Right to Refuse or Withdraw

You do not have to take part in this research if you do not wish to do so. You may also stop participating in the research at any time you choose. It is your choice and all of your rights will still be respected.

Alternatives to Participating

If you do not wish to take part in the research, you will be provided with the established standard treatment available at the center/institute/hospital. People who have malaria are given

DETAILED DESCRIPTION:
Detailed Description This research project, titled "Prophylactic IV paracetamol in extremely premature infants: A Palestinian-Based Study," aims to investigate the efficacy of prophylactic intravenous paracetamol in preventing Patent Ductus Arteriosus (PDA) in extremely premature infants born at less than 30 weeks of gestation or with a birth weight below 1250 grams. The study will be conducted in Palestine Medical Complex, Al Makassed,and Al Ahli hospitals.

Background:

Patent Ductus Arteriosus (PDA) is a common cardiovascular complication in premature and low birth-weight infants. While it typically closes spontaneously in full-term infants, it often remains open in premature infants, leading to hemodynamically significant PDA (HSPDA) with potential cardiopulmonary distress. Current pharmacological interventions to promote PDA closure include NSAIDs like indomethacin and ibuprofen, which carry risks of adverse effects such as renal impairment and gastrointestinal complications. Paracetamol has emerged as a potential alternative due to its cyclooxygenase (COX) inhibitory effects and a potentially safer profile. This study seeks to evaluate the effectiveness of prophylactic IV paracetamol in reducing the incidence of PDA and its associated complications in this vulnerable population.

Study Design:

This is a prospective, double blinded randomized controlled clinical trial. The study will compare the incidence of PDA requiring medical or surgical intervention, as well as various short-term and long-term neonatal outcomes, between a group receiving prophylactic IV paracetamol and a control group.

Method of randomisation: The randomisation will be done using envelopes which are labeled as "give paracetamol" or "don't give paracetamol". Each participant will be assigned to a random envelop and will be given or not given the intervention without the researchers or the participant knowing if they received the IV prophylactic paracetamol.

Intervention:

The intervention involves the prophylactic administration of intravenous paracetamol to extremely premature infants. The specific dosage and duration of paracetamol administration will be detailed in the full protocol.

Participant Population:

The study will enroll inborn babies with gestational ages of less than 30 weeks or birth weight below 1250 grams. Participants will be recruited from Palestine Medical Complex, Al Makassed, and Al Ahli hospitals.

Data Collection and Management:

Data will be collected using a standardized data sheet. This sheet includes variables such as:

Patient ID Gender Date of birth Weeks of gestation Echocardiography findings at 72 hours after birth and during long-term follow-up (PDA presence, size, transductal diameter) Presence of other outcomes (Mortality, Bronchopulmonary dysplasia, Severity of respiratory distress syndrome, Definitive sepsis, Massive pulmonary hemorrhage, Intraventricular hemorrhage, Oxygen requirements at 28 days postnatal age, Necrotizing enterocolitis, Retinopathy of prematurity, Neurodevelopmental disorders, Growth retardation) AST & ALT levels at 24 hours and 72 hours after course completion.

Ethical Considerations:

The study protocol, consent form, and data sheet have been prepared in accordance with ethical guidelines. Informed consent will be obtained from the parents or legal guardians of the eligible infants. The consent form clearly outlines the purpose of the research, procedures, potential risks (including known side effects of paracetamol therapy), and benefits. Participants will be assured of their right to withdraw from the study at any time without penalty. The application form indicates potential risks to participants include physical harm, physical discomfort, psychological/emotional harm, psychological/emotional discomfort, and legal repercussions. Risk management procedures include addressing known side effects of FDA-approved paracetamol therapy. The study has been submitted for approval by the Al-Quds University Research Ethics Committee.

Statistical Analysis Plan:

The statistical analysis plan will describe the methods used to analyze the collected data to address the primary and secondary objectives. This will likely involve comparing the incidence of PDA and other outcomes between the intervention and control groups using appropriate statistical tests (e.g., chi-square test for categorical variables, t-tests or non-parametric tests for continuous variables). Time-to-event analysis may be used for outcomes like PDA closure. Subgroup analyses may be performed based on gestational age, birth weight, or other relevant factors. The plan will also address methods for handling missing data and potential confounders.

Quality Assurance and Data Validation:

Data validation will involve double-checking entered data against source documents (medical records). Data checks will be implemented to identify inconsistencies or out-of-range values. Regular monitoring of data collection procedures will ensure accuracy and completeness.

Sample Size Assessment:

The proposal references several studies and indicates that previous research suggests paracetamol may accelerate PDA closure. A formal sample size calculation was performed to determine the number of participants required to detect a statistically significant difference in the primary outcome measure, for a significance level of 0.05, and a power of 0.8 and considering the sample size treat/control ratio to be 0.05, the total sample size was calculated to be 28.

Research Personnel:

The principal investigators are Dr. Hadeel Atout and Dr. Mohammed Khwaira from Al-Quds University. Dr. Sarah Alkhatib is the mentor, and the students involved are Yasmeen Jaber, Adham Qadamani, Amro Sinokrot, Fares Sayed Ahmad, Issa Mansour, and Nidal Muna.

ELIGIBILITY:
Inclusion Criteria:

* gestational ages of <30 weeks or birth weight below 1250 gm
* inborn babies
* authorization to perform the study signed by one of the parents after receiving enough information about the condition

Exclusion Criteria:

* Outborn babies
* The presence of a significant birth defect or a congenital anomaly
* Clinical instability that can lead to rapid death

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Presence of patent ductus arteriosus | 72 hours
  The primary outcome is the presence of patent ductus arteriosus (diagnosed by echocardiography)

SECONDARY OUTCOMES:
mortality | Within 1 month of birth
bronchopulmonary dysplasia | 36 weeks corrected gestational age
  bronchopulmonary dysplasia (diagnosed as the participant still needing oxygen requirements at 36 weeks corrected gestational age)
severity of respiratory distress syndrome | Within 1 month of birth
  defined as use of more than two doses of surfactant
Definitive sepsis | Within 1 month of birth
  (clinical symptoms and signs of sepsis and a positive bacterial blood culture in a specimen obtained by sterile technique
Massive pulmonary hemorrhage | Within 1 month of birth
Intraventricular hemorrhage (grade III or IV) | Within 1 month of birth
oxygen requirements at 28 days postnatal age | 28 days after birth
necrotizing enterocolitis (stage 2 or 3) | Within 1 month of birth
Retinopathy of prematurity | 4-9 weeks after birth
Liver enzymes | at 24 hours, and at 72 hours of birth, in addition to after completion of the paracetamol course
  AST and ALT

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel Atout, MD, Principal Investigator — Palestine Medical Complex and Al-Quds University.
Locations (3):
- Palestinian Territories (3):
  - Makassed, East Jerusalem
  - Al Ahli Hospital, Hebron
  - Palestine Medical Complex, Ramallah